CLINICAL TRIAL: NCT04878276
Title: Randomised, Investigator-blinded, Controlled, Multicentre Comparative Study on the Treatment of Head Lice Infestation With 2 Dimeticone Preparations With Different Application Times and Compositions: Dimet 5® (100% Dimeticon) Versus Hedrin® Once Liquid Gel (4% Dimeticon + Nerolidol)
Brief Title: Comparative Head Lice Therapy With Dimet 5® vs. Hedrin® Once
Acronym: VEKODIH
Status: Recruiting | Type: Observational
Sponsor: Infectopharm Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: VEKODIH
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Head Lice Infestation; Pediculosis Capitis; Lice
MeSH Terms: conditions — Lice Infestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dimet 5: Dimet 5 is a certified medical device for the treatment of head lice infestation. It contains only ("liquid") dimeticone oil and, when used correctly, enables physical killing of head lice and their eggs.
  Interventions: Device: Dimet 5
- Hedrin Once Liquid Gel: Hedrin Once Liquid Gel is a certified medical product for the removal of head lice and nits. The liquid gel contains 4% dimethicone and nerolidol (Penetrol®).
  Interventions: Device: Dimet 5

INTERVENTIONS:
Device: Dimet 5 — The application is carried out according to the enclosed instructions for use.

SUMMARY:
Randomized, investigator-blinded, controlled, multicenter comparative study on the treatment of acute head lice infestation in children with 2 dimeticone preparations with different application times and compositions: Dimet 5® (100% dimeticone) versus Hedrin® Once Liquid Gel (4% dimeticone + nerolidol) with treatment success assessment via freedom from infestation of live head lice at final examination at V2, i.e. day 19 after first treatment.

ELIGIBILITY:
Inclusion Criteria:

* Acute head lice infestation
* Age ≥ 6 months
* Adequate informed consent for study participation:

  * Age-appropriate informed consent and verbal informed consent from the patient (if capable of both).
  * Written informed consent from the legal guardian(s) (written and verbal).

Exclusion Criteria:

* Adults (≥ 18 years of age)
* Known hypersensitivity to any component of the test or comparator product.
* Scalp lice therapy in the previous 2 weeks (with an appropriate drug or medical device).
* Severe disease of the scalp or injuries/open wounds on the hairy head
* Secondary infection in the area of the hairy head
* Treatment with cotrimoxazole or trimethoprim in the last 4 weeks or new treatment to be initiated now
* Other relevant reasons, e.g. diseases or dysfunctions, which, in the opinion of the investigator, militate against the inclusion of the patient in the study (including risk factors for severe COVID-19 disease in the case of SARS-CoV-2 infection)
* Simultaneous participation of another household member in the trial.
* Previous participation in this trial
* Participation in another trial within the last 30 days
* Inability of the legal guardian(s) to understand the study content and instructions.
* Limited legal capacity of the legal guardian(s)
* Apparent unreliability or unwillingness to cooperate on the part of the legal guardian(s)
* Known alcohol, medication or drug dependency of the legal guardian(s)
* Dependence of the patient or guardian on the sponsor or investigator.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children ≥ 6 months with acute head lice infestation
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Freedom from infestation | Day 17 to 21
  Freedom from infestation of live head lice at the final examination (V2)

CONTACTS AND LOCATIONS:
Locations (26):
- Germany (26):
  - Dr. med. Thilo Heising, Aalen
  - Gemeinschaftspraxis Gilb/Bauer/von Bentzel, Augsburg
  - Dr. med. Omar Esteban Fernandez Salgueiro, Balingen
  - Dr. med. Martin Wiesner, Berlin
  - Praxis für Kinder- und Jugendheilkunde, Blankenfelde
  - Gemeinschaftspraxis für Kinder- und Jugendmedizin, Bremen
  - Kinderarztpraxis Vaitl, Chemnitz
  - Praxis Dr. Glatzel, Düsseldorf
  - Kinderarztpraxis Dr. Lichtenstein, Eschborn
  - Kinderarztpraxis Dr. Zumegen, Essen
  - Kinderärztliche Gemeinschaftspraxis Tost/Lange, Greifswald
  - Gemeinschaftspraxis Dreher/Hübler, Guelders
  - Dr. med. Friedrich Kaiser, Hamburg
  - Dr. med. Ludwig Stapenhorst, Hürth
  - Kinderarztpraxis Dr. Hable, Leipzig
  - Kinderärzte im Karree, Leverkusen
  - Dr. med. Susanne Ludwig, Lübeck
  - Kinderarztpraxis Dr. Bach, Mainz
  - Dr. med. Katrin Biebach, München
  - Kinderarztpraxis am Ringmarkt, Neuwied
  - Giraffenpraxis, Ratingen
  - Kinderarztpraxis Dr. Steinmetz, Saarbrücken
  - Kinderarztpraxis Dr. Klink, Schwarzenberg
  - Simon Traub, Schweigen-Rechtenbach
  - Kinder- und Jugendarztpraxis, Weil am Rhein
  - PediaMed Wolfsburg, Wolfsburg

IPD SHARING:
Plan to Share IPD: No